CLINICAL TRIAL: NCT04731766
Title: Effectiveness of Using Nano-Silver Fluoride Varnish Versus Sodium Fluoride Varnish in Management of Cervical Dentin Hypersensitivity in Adult Patients: A Randomized Clinical Trial.
Brief Title: Effect of Using Different Varnishes on Dentin Hypersensitivity; Na Fluoride and Nano-silver Fluoride
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nayera Hassanien Mohamed (Other)
Responsible Party: Sponsor-Investigator, Nayera Hassanien Mohamed, Assistant Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205
Record Dates: First submitted 2020-10-06; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrine 5% Sodium Fluoride (Active Comparator): It was developed to prolong the contact between the tooth surface and fluoride to increase the resistance against caries attack and manage tooth hypersensitivity; the active ingredient of fluoride varnish is mostly 5% sodium fluoride.
  Interventions: Behavioral: Citrine 5 % sodium fluoride
- concocuted Nano-silver fluoride (Experimental): Nano-silver fluoride (NSF) is a laboratory synthesized solution
  Interventions: Behavioral: concocted nano-silver fluoride

INTERVENTIONS:
Behavioral: Citrine 5 % sodium fluoride — Citrine varnish is a 5% sodium fluoride varnish, It was developed to prolong the contact between the tooth surface and fluoride to increase the resistance against caries attack and manage tooth hypersensitivity; the active ingredient of fluoride varnish is mostly 5% sodium fluoride.
  Arms: Citrine 5% Sodium Fluoride
Behavioral: concocted nano-silver fluoride — Nano-silver fluoride (NSF) is a solution which has been introduced as an experimental formulation in which it's stability for three years has been proved by Santos et al. The laboratory synthesis of concocted NSF was carried out in a nano-technology center; Several trials were done until we have reached a successful end product.
  Arms: concocuted Nano-silver fluoride

SUMMARY:
2 different varnishes will be used to test their effectiveness in controlling teeth hypersensitivity in adult patient.

DETAILED DESCRIPTION:
In-vivo part:

Each varnish will be applied separately on different teeth according to the manufacturer's instructions and the VAS will be measured according to a specific timeline: T0 (baseline, before application of varnish), T1 (1 week after application), T2 (4 weeks after application) and T3 (4 weeks after application).

In-situ part:

Dentin specimen will be prepared from extracted teeth from the orthodontic department in our college, sterilized and prepared.

it will be bonded to an orthodontic wire and bonded to upper first molar. Dentinal occlusion will be measured using scanning electron microscope following the same timeline.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting in one of the Qasr Einy, faculty of dentistry outpatient clinics.
* Males or females.
* Patient's age range 25-50 years.
* Patients complaining of hypersensitive areas on facial surfaces of the teeth (incisors, cuspids, bi-cuspids, and first molars with exposed cervical dentine) with teeth scoring Bpain (VAS score: greater than or equal to 3) during application of stimulus (airblast and tactile sensitivity test).
* Tooth with exposed root surface, complaining from hypersensitivity (VAS score; greater than or equal to 3).
* Patients accept the 2-months follow-up period.
* Provide informed consent.

Exclusion Criteria:

* • Patients participating in another dental study that may alter the results of this study.

  * A medical condition that could hinder the accuracy of pain reporting (e.g., pain disorders).
  * Any chronic medical condition that requires the regular use of anti-inflammatory pain medications.
  * Patients used or applied a desensitizing varnish within the last four weeks.
  * Patients with dental problems; chipped teeth, defective restorations, fractured Un-displaced cuspids or deep dental caries.
  * Lack of patient's approval and compliance.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
change in dentin Hypersensitivity | 1 week, 4 weeks & 8 weeks
  Visual Analogue Scale (VAS) will be used; 0 is no pain and 10 is severe pain. Pictures are added to the same, as well as colors to guide the patient during selection of pain severity.

SECONDARY OUTCOMES:
change in dentinal Tubule Occlusion | 1 week, 4 weeks * 8 weeks
  the dentinal tubule occlusion of citrine 5% sodium fluoride and the dentinal tubule occlusion of nano-silver fluoride for treatment of dentin hypersensitivity and compare them together

IPD SHARING:
Plan to Share IPD: No